CLINICAL TRIAL: NCT00720460
Title: Technical Development of Interventional Cardiovascular Magnetic Resonance Imaging in Healthy Volunteers
Brief Title: Technical Development of Interventional Cardiovascular Magnetic Resonance Imaging in Normal Volunteers
Status: Terminated | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080185; 08-H-0185
Record Dates: First submitted 2008-07-19; First posted 2008-07-22 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2018-11-02

CONDITIONS: Healthy
Keywords: Magnetic Resonance Imaging; Minimally Invasive Therapy; Transcatheter Therapeutics; Healthy Volunteers; Gadolinium Contrast; Healthy Volunteer; HV

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Experimental: Healthy Volunteers

SUMMARY:
This study will test new techniques to image the heart, blood vessels, and legs using magnetic resonance imaging (MRI). The techniques will be used to plan and guide treatments using minimally invasive methods.

Healthy normal volunteers 18 years of age and older may be eligible for this study.

For MRI, the subject lies flat on a table that can slide in and out of the scanner, a metal cyclinder. Special antennas, covered in pads, are placed against the subject s body. The scan time can vary from 20 minutes to 2 hours, with most scans lasting between 45 and 90 minutes. The subject may be asked to wear adhesive patches on the chest for monitoring the heart and a belt or finger pad for monitoring breathing. During the test, a contrast agent called gadolinium may be injected. This substance brightens the heart and arteries during the scan, providing a better picture of blood flow.

During the procedure, subjects may be asked to exercise their legs on a machine to evaluate the effects of motion and exercise on the MRI exam.

Large blood pressures cuffs may be placed on either or both thighs or calves to try to measure arterial flow to the legs. The cuffs are inflated to a pressure as high as at least 50 mmHg higher than thesubject s systolic blood pressure (up to 250 mmHg) for up to 10 minutes.

Subjects may be asked to return for repeated scans.

DETAILED DESCRIPTION:
We will evaluate new developments in fast magnetic resonance imaging (MRI) of the heart and blood vessels on healthy volunteers. These studies will be conducted in the NIH MRI systems located at the NIH Clinical Center in Bethesda, Maryland. These procedures may involve the intravenous administration of commercially available MR contrast media, supine exercise or the inflation of blood pressure cuffs on the lower extremities during the MRI imaging. The results will be used to evaluate the performance of various research pulse sequences, gradient coils, and radiofrequency receiver coils on human subjects and will provide essential ground work for specific patient protocols, both diagnostic and therapeutic.

ELIGIBILITY:
* 1. GENERAL INCLUSION CRITERIA:
* Healthy adult volunteers, age is greater than 18 years of age, who consent to participate in writing

  2. EXCLUSION CRITERIA: MRI risk
* Cardiac pacemaker or implantable defibrillator
* Cerebral aneurysm clip
* Implanted neural stimulator (e.g. TENS-Unit)
* Any type of ear or cochlear implant
* Intra-ocular foreign body (e.g. metal shavings)
* Any implanted device (e.g. insulin pump, drug infusion device)
* Metal shrapnel or bullet
* Morbid obesity
* Claustrophobia

  3. EXCLUSION CRITERIA: Contrast media risk:
* Pregnant women (when uncertain, subjects will undergo urine or blood testing) or lactating women
* Known hemoglobinopathy
* Known kidney disease
* Exposure to gadolinium MRI contrast agents in the past 18 hours, if the study requires gadolinium MRI contrast agent.
* Diabetes
* Children are not included.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2008-07-18; Study Completion 2018-11-02

PRIMARY OUTCOMES:
To develop and test new and incremental approaches to fast cardiovascular MRI in healthy human subjects. (healthy volunteers) | Day of study
  There are 24 objectives listed in the protocol as potential outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Lederman, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Lederman RJ. Cardiovascular interventional magnetic resonance imaging. Circulation. 2005 Nov 8;112(19):3009-17. doi: 10.1161/CIRCULATIONAHA.104.531368. No abstract available. PMID 16275886
- [Background] Haustein J, Laniado M, Niendorf HP, Louton T, Beck W, Planitzer J, Schoffel M, Reiser M, Kaiser W, Schorner W, et al. Triple-dose versus standard-dose gadopentetate dimeglumine: a randomized study in 199 patients. Radiology. 1993 Mar;186(3):855-60. doi: 10.1148/radiology.186.3.8430199.
- [Background] Niendorf HP, Haustein J, Cornelius I, Alhassan A, Clauss W. Safety of gadolinium-DTPA: extended clinical experience. Magn Reson Med. 1991 Dec;22(2):222-8; discussion 229-32. doi: 10.1002/mrm.1910220212. PMID 1812350
- [Derived] Saybasili H, Kellman P, Griswold MA, Derbyshire JA, Guttman MA. HTGRAPPA: real-time B1-weighted image domain TGRAPPA reconstruction. Magn Reson Med. 2009 Jun;61(6):1425-33. doi: 10.1002/mrm.21922. PMID 19353673